CLINICAL TRIAL: NCT07339527
Title: An Open-label, Multicenter, Exploratory Clinical Study of the EZH2 Inhibitor Zeprumetostat in Combination Therapy for Patients With Relapsed or Refractory Mature T-cell and NK-cell Lymphomas.
Brief Title: EZH2 Inhibitor Zeprumetostat in Combination Therapy for Patients With Relapsed or Refractory Mature T-cell and NK-cell Lymphomas
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-804
Record Dates: First submitted 2025-12-20; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Mature T-cell and NK-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zeprumetostat Combined with Golidocitinib or Chidamide (Experimental): In Cohort 1, patients will receive Zeprumetostat in combination with Golidocitinib, with an initial dose of 350mg of Zeprumetostat. Each treatment cycle is 28 days. The Zeprumetostat will be combined with Golidocitinib at the RP2D dose level for an extension study. In Cohort 2, patients will receive Zeprumetostat in combination with Chidamide, with an initial dose of 350mg of Zeprumetostat. Each treatment cycle is 28 days. The Zeprumetostat will be combined with Chidamide at the RP2D dose level for an extension study.
  Interventions: Drug: Zeprumetostat; Drug: Golidocitinib; Drug: Chidamide

INTERVENTIONS:
Drug: Zeprumetostat — 350mg, po, bid
Drug: Golidocitinib — Cohort 1: Golidocitinib: 150mg, po, qd
Drug: Chidamide — Cohort 2: Chidamide: 20mg, po, biw

SUMMARY:
This is a prospective, multicenter, open-label, phase Ib/II clinical study to evaluate the safety and efficacy of EZH2 inhibitor Zeprumetostat in combination therapy for patients with relapsed or refractory mature T-cell and NK-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study; fully understand and be informed about the study and sign the Informed Consent Form (ICF); willing to comply with and capable of completing all trial procedures;
* Age ≥ 18 years
* Pathologically confirmed mature T-cell and NK-cell lymphomas.
* Using the Lugano 2014 criteria, the patient must have at least one measurable or evaluable lesion
* Participants must have experienced disease progression, treatment failure, or intolerance following standard therapy. Patients with ALCL are required to have previously received anti-CD30-targeted therapy, while patients with NKTCL must have previously been treated with pegaspargase or L-asparaginase.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ and bone marrow function

Exclusion Criteria:

* Lymphoma involvement in the central nervous system or meninges
* Active infections
* Prior treatment with an EZH2 inhibitor or an EZH1/2 dual inhibitor that was discontinued due to intolerance to toxicity;
* For patients enrolled in Cohort 1, prior treatment with a JAK inhibitor that was discontinued due to intolerance to toxicity;
* For patients enrolled in Cohort 2, prior treatment with an HDAC inhibitor that was discontinued due to intolerance to toxicity.
* History of Human Immunodeficiency Virus (HIV) infection and/or Acquired Immunodeficiency Syndrome (AIDS).
* Patients with mental disorders or those unable to provide informed consent
* Any other condition deemed by the investigator to be unsuitable for study enrollment;
* Pregnant or breastfeeding women, and subjects of childbearing potential who are unwilling to use contraception;
* Individuals with a known hypersensitivity to any of the investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
DLT for Phase 1b | The first cycle after administration (each cycle is 28 days)
  To identify the dose-limiting toxicity
Overall response rate(ORR) for Phase 2 | Up to 24 months
  The proportion of patients who achieve complete remission (CR) or partial remission (PR) as the best response.
RP2D for phase Ib | The first cycle after administration (each cycle is 28 days)
  To identify the recommended phase 2 dose

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to 24 months
  Defined as the proportion of patients who achieve complete remission as the best response
Duration of Response(DOR) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Progression-free survival(PFS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy
Overall survival(OS) | Up to 4 years
  To investigate the preliminary anti-tumor efficacy

IPD SHARING:
Plan to Share IPD: Undecided